CLINICAL TRIAL: NCT04575181
Title: A Multiple Dose, Randomised, Double Blinded, Double Dummy Trial Investigating Efficacy and Safety of NNC0268-0965 Versus Insulin Glargine in Subjects With Type 2 Diabetes Mellitus
Brief Title: A Clinical Study to Compare the Efficacy and Safety of a Novel Medicine (NNC0268-0965) With Insulin Glargine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN1965-4485; U1111-1243-0598 (Other: World Health Organization (WHO)); 2019-004381-18 (Registry Identifier: European Medicines Agency (EudraCT))
Record Dates: First submitted 2020-09-28; First posted 2020-10-05 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- NNC0286-0965 (Experimental): NNC0286-0965 administered together with insulin glargine placebo. If previously treated with oral anti-diabetic drugs (OADs), participants will remain on these in the trial
  Interventions: Drug: NNC0268-0965; Drug: Placebo (insulin glargine)
- Insulin glargine (Active Comparator): Insulin glargine administered together with NNC0286-0965 placebo. If previously treated with OADs, participants will remain on these in the trial
  Interventions: Drug: Insulin glargine; Drug: Placebo (NNC0268-0965)

INTERVENTIONS:
Drug: NNC0268-0965 — For subcutaneous (s.c., under the skin) injection once daily for 26 weeks
  Arms: NNC0286-0965
Drug: Insulin glargine — For s.c. injection once daily for 26 weeks
  Arms: Insulin glargine
Drug: Placebo (NNC0268-0965) — For s.c. injection once daily for 26 weeks
  Arms: Insulin glargine
Drug: Placebo (insulin glargine) — For s.c. injection once daily for 26 weeks
  Arms: NNC0286-0965

SUMMARY:
The study will look at the efficacy and safety of NNC0268-0965 (referred to as insulin 965). The study aims to show that insulin 965 has positive effects on the blood vessels. Participants will get either the new insulin 965 or insulin glargine - a medicine that doctors already can prescribe (Lantus®). Which treatment participants get is decided by chance. Participants will self-administer 2 injections per day under the skin of the thighs for 26 weeks. Study participation will last for about 32 weeks. Participants will have 15 clinic visits, 2 magnetic resonance imaging (MRI) visits and 14 phone calls with the study doctor. There will be a number of in-house assessments to study the effect of the new insulin. The assessments will be explained later in detail. The treatment of disease is not an aim of this study. Participants cannot be in the study if the study doctor thinks that there are risks for their health. Women can only take part in the study if they are not able to become pregnant.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial related activities. Trial related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial.
* Aged 40-75 years (both inclusive) at the time of signing informed consent.
* Diagnosed with diabetes mellitus, type 2 (T2DM) at least 180 days prior to the day of screening.
* Male subject or female subject of non-childbearing potential. Non-childbearing potential being surgically sterilised (i.e. documented hysterectomy, bilateral salpingectomy or bilateral oophorectomy or being postmenopausal (as defined as no menses for 12 months without an alternative medical cause) prior to the day of screening.
* HbA1c at screening between 6.0 and 10.0%, both inclusive.
* Treated with or without any oral antidiabetic agents including any metformin formulations, dipeptidyl peptidase 4 (DPP-4) inhibitors, Sodium-glucose co-transporter-2 (SGLT-2) inhibitors, alpha glucosidase inhibitors, sulfonylureas (including meglitinides). If treated with oral antidiabetic agents, the total daily dose must have been stable within the past 30 days prior to the day of screening.
* Treated with basal insulin regimen at least 90 days prior to the day of screening with a total daily dose of:
* equal to or above 10U/day if HbA1c above 7.5%
* equal to or above 15U/day if HbA1c above 6.5% and equal to or below 7.5%
* equal to or above 25U/day if HbA1c equal to or below 6.5%

Exclusion Criteria:

* Previous exposure to insulin 287 formulation A (i.e. trial NN1436-4057).
* Any of the following which in the investigator's opinion might jeopardise subject's safety or interfere in relation to the magnetic resonance scans: metallic implants, pacemaker, defibrillator, artificial valves in heart, internal electrical devices (e.g. cochlear implant, nerve stimulator, brain stimulator, gastric pacemaker, bladder stimulator etc.) magnetic clips, confirmed claustrophobia or permanent makeup, working or has worked as a metal worker or welder.

Note: Up to 18 subjects, who are not able to have the MRI scan performed, will be allowed inclusion, at the investigator's discretion.

-. Myocardial infarction, stroke, hospitalisation for unstable angina pectoris or transient ischaemic attack within 180 days to the day of screening.

* Presently classified as being in New York Heart Association (NYHA) Class III or IV.
* Renal impairment measured as an Estimated Glomerular Filtration Rate (eGFR) value of below 45.0 mL/min/1.73 m^2 as defined by Kidney Disease Improving Global Outcomes (KDIGO) 2012 at screening.
* Recurrent severe hypoglycaemic episodes within the last year as judged by the investigator.
* Inadequately treated BP defined as Grade 3 hypertension or higher (Systolic equal to or above 160 mmHg or diastolic equal to or a bove 100 mmHg) at screening based upon mean blood pressure of the last 2 of 3 measurements.
* Treatment with any medication for the indication of diabetes or obesity other than stated in the inclusion criteria within the past 30 days or 5 times the half-life of the product, whichever timeframe is longest prior to the day of screening.
* Planned initiation of concomitant medications known to affect weight or glucose metabolism (e.g. treatment with orlistat, thyroid hormones, or systemically effective corticosteroids).
* Use of statins (unless the use of these has been stable during the past 3 months) or use of systemically effective corticosteroids, monoamine oxidase (MAO) inhibitors, systemic non-selective beta-blockers, growth hormone, non-routine vitamins or herbal products at screening.
* Rotating or permanent night shift worker.
* Uncontrolled and potentially unstable diabetic retinopathy or maculopathy. Verified by a fundus examination performed within the past 90 days prior to screening or in the period between screening and randomisation. Pharmacological pupil-dilation is a requirement unless using a digital fundus photography camera specified for non-dilated examination.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2021-12-24 (Actual)

PRIMARY OUTCOMES:
Change in flow mediated dilation | From Visit 3B (week 0) to visit 30B (week 26)
  Percent

SECONDARY OUTCOMES:
Change in pulse wave velocity | From Visit 3B (week 0) to visit 30B (week 26)
  m/s
Change in leg blood flow | From Visit 3B (week 0) to visit 30B (week 26)
  ml/100 ml/min
Change in retinal arteriolar dilation | From Visit 3A (week 0) to visit 30A (week
  Percent
Relative change in liver fat percentage measured by magnetic resonance imaging proton density fat fraction (MRI-PDFF) | From Visit 2 (week 0) to visit 29 (week 26)
  Ratio
Change in left ventricular ejection fraction | From Visit 2 (week 0) to visit 29 (week 26)
  Percent
Change in glycosylated haemoglobin (HbA1c ) | From Visit 3B (week 0) to visit 30B (week 26)
  Percent
Change in body weight | From Visit 3B (week 0) to visit 30B (week 26)
  kg
Change in body fat mass as measured by BOD POD (a method for determining the lean body mass) | From Visit 3B (week 0) to visit 30B (week 26)
  Percent
Relative change in rate of glucose disposal at short Insulin Tolerance Test | From Visit 3B (week 0) to visit 30B (week 26)
  Ratio
Number of adverse events | From Visit 3B (week 0) to visit 30B (week 26)
  Number of events
Number of severe hypoglycaemic episodes (level 3) | From Visit 3B (week 0) to visit 30B (week 26)
  Number of episodes
Number of clinically significant hypoglycaemic episodes (level 2) (below 3.0 mmol/L (54 mg/dL), confirmed by BG meter) or severe hypoglycaemic episodes (level 3) | From Visit 3B (week 0) to visit 30B (week 26)
  Number of episodes
Number of clinically significant hypoglycaemic episodes s (level 2) ((below 3.0 mmol/L (54 mg/dL), confirmed by BG meter) | From Visit 3B (week 0) to visit 30B (week 26)
  Number of episodes

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (1452), Study Director — Novo Nordisk A/S
Locations (2):
- Germany (2):
  - Profil GmbH & Co. KG, Mainz
  - Profil Institut für Stoffwechselforschung GmbH, Neuss

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com